CLINICAL TRIAL: NCT04472884
Title: mWACh-PrEP: A SMS-based Support Intervention to Enhance PrEP Adherence During Pregnancy and Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); Jomo Kenyatta University of Agriculture and Technology (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jillian Pintye, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010797; 1R01NR019220-01A1 (NIH)
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: HIV Infections; Pregnancy Related; Adherence, Medication
Keywords: pre-exposure prophylaxis; HIV prevention; PrEP
MeSH Terms: conditions — HIV Infections; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mWACh-PrEP (Experimental)
  Interventions: Behavioral: mWACh-PrEP; Other: Standard of Care
- Standard of Care (Other)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: mWACh-PrEP — Participants randomized to mWACh-PrEP will be registered into the system, in addition to receipt of SOC services. Women registered into the mWACh-PrEP platform will indicate their preferences for message delivery including a preferred name for messaging, language (English or Kiswahili or Dholuo), and day of the week and time for SMS delivery. Once registered, women will receive weekly automated push messages on the day/time of their choice from enrollment through 6-months postpartum. All automated push messages will include participant nickname, clinic and nurse name, an educational message or actionable advice targeting PrEP adherence and continuation and/or maternal and child health (MCH) topics, and a question related to the content. SMS topics will include adherence encouragement, PrEP efficacy and safety, self-efficacy for prevention of HIV, support for potential PrEP side effects, behavioral skills (tips for remembering PrEP medications) and visit reminders.
  Arms: mWACh-PrEP
Other: Standard of Care — All participants will receive SOC services for MCH and PrEP that will include health education, clinical assessments, laboratory safety monitoring, STI (syphilis, gonorrhea, and chlamydia) screening and treatment (including expedited partner treatment for

SUMMARY:
In high HIV prevalence regions, women are at high risk for HIV during pregnancy and breastfeeding. To protect women and reach elimination of mother-to-child HIV transmission, the World Health Organization recommends offering oral tenofovir (TFV)-based pre-exposure prophylaxis (PrEP) to HIV-negative pregnant and postpartum women in high-burden settings. Although most pregnant Kenyan women with HIV risk factors accept PrEP when offered, >50% discontinue PrEP within 30 days of initiation and sub-optimal adherence is common. To date, no intervention studies to improve PrEP adherence include pregnant or postpartum women. The investigators adapted an SMS communication platform (mWACh) to send PrEP-tailored, theory-based SMS to facilitate adherence among pregnant women who initiate PrEP. In a non-randomized pilot, the investigators found that mWACh-PrEP recipients were more likely to persist with PrEP use and to self-report high adherence. The investigators propose a randomized trial to determine the effect of the mWACh-PrEP tool on PrEP adherence during pregnancy through the postpartum period. The investigators will also gather data on cost and delivery using the Proctor Implementation Outcomes Framework to expedite translation into routine practice. The overarching hypothesis is that mWACh-PrEP will improve PrEP adherence among mothers at-risk for HIV, be acceptable to patients and providers, and be cost-effective. The study will be executed via the following aims:

Aim 1- To determine the effect of the mWACh-PrEP tool on PrEP adherence during pregnancy through the postpartum period among women who initiate PrEP within ANC-PrEP. We will conduct a 2-arm randomized trial comparing mWACh-PrEP vs standard of care (SOC, i.e. in-clinic adherence counseling) among HIV-uninfected pregnant women with high HIV acquisition risk (defined by validated risk score) who initiate PrEP. The primary outcome will be adherence at 6 months postpartum (TFV hair levels >0.038 ng/mg; consistent with 7 pills/ week). Secondary outcomes will include sexually transmitted infection (STI) incidence, adherence cofactors, and prevention-effective adherence (time-varying alignment of adherence with risk behaviors). Exploratory outcomes will include HIV incidence and perinatal outcomes by arm. Hypothesis: mWACh-PrEP will increase PrEP adherence compared to SOC.

Aim 2- Evaluate barriers and facilitators of mWACh-PrEP implementation within routine ANC. Using the Proctor framework, we assess acceptability and feasibility by conducting interviews and focus-groups with ANC-PrEP users, providers, and health planners. Hypothesis: Indications for readiness of mWACh-PrEP will be identified.

Aim 3- Estimate the cost-effectiveness of implementing mWACh-PrEP within ANC-PrEP, per HIV infection and disability-adjusted life-year (DALY) averted. We use data from Aims 1 and conduct micro-costing and time-and-motion studies to estimate the cost of mWACh-PrEP from a payer perspective. The incremental cost-effectiveness ratio (ICER) per HIV infection and DALY averted compared to SOC will be calculated. Hypothesis: Incorporating data on PrEP and ANC outcomes with improve ICERs for mWACh-PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting for routine antenatal care (ANC) who are:
* ≥18 years old
* 24-32 weeks gestation
* No documented tuberculosis infection
* HIV negative (based on ANC HIV testing)
* Plan to reside in area for at least one year postpartum
* Plan to receive antenatal, postnatal, and infant care at study facility
* Initiated PrEP during routine ANC
* Have an HIV risk score >6 (based on Pintye et al 2017).

Exclusion Criteria:

* Do not plan to remain in the study site catchment area for at least 1 year
* Do not have mobile phones.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
% of participants with detectable TFV levels in hair >0.038 ng/mg (PrEP adherence) | 6-months postpartum
  PrEP adherence will be measured with a binary endpoint (Yes/No) based on hair samples from 6-month postpartum visits. Detectable TFV levels in hair >0.038 ng/mg (consistent with 7 doses/week) will be considered adherent. If a participant stopped PrEP use or exited the study before 6 months postpartum (ie had no hair sample collected), the participant will be considered non-adherent

SECONDARY OUTCOMES:
% of participants with detectable TFV levels in hair >0.038 ng/mg (Sustained PrEP adherence) | 9-months postpartum
  Binary endpoint (Yes/No) of detectable TFV levels in hair >0.038 ng/mg (consistent with 7 doses/week) at 9-months postpartum (3 months after cessation of mWACh messaging). Same definition of non-adherence as above.
% of participants with <90% PrEP adherence or discontinuation (Predictors of non-adherence) | 6-months postpartum
  Factors associated with poor adherence (outcomes of <90% adherent on PrEP or discontinuation) will include demographics, relationship/partner characteristics, psychosocial factors, socioeconomic status, low health/HIV literacy, fear of disclosure
Incidence of STI diagnoses | 6-months postpartum
  Frequency of STI (syphilis, gonorrhea, chlamydia) detection at follow-up visits will be compared between randomization arms

OTHER OUTCOMES:
Incidence of HIV acquisition | 6-months postpartum
  Frequency of HIV diagnosis at follow-up visits will be compared between randomization arms
% of participants who experience preterm birth, neonatal death, and infant growth faltering | 6-months postpartum
  Frequency of preterm birth, neonatal death, and infant growth faltering outcomes will be compared between randomization arms
% of participants who offer male partners expedited partner therapy (EPT) | 6-months postpartum
  Among women with STI diagnoses, frequency of offering male partners EPT will be compared between randomization arm

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Pintye, RN, MPH, PhD, Principal Investigator — University of Washington
Locations (4):
- Kenya (4):
  - Kisumu County Referral Hospital, Kisumu
  - Lumumba Sub County Hospital, Kisumu
  - Migosi Sub County Hospital, Kisumu
  - Yala Sub County Hospital, Siaya

REFERENCES:
- [Derived] Mogaka JN, Otieno FA, Akim E, Beima-Sofie K, Dettinger J, Gomez L, Marwa M, Odhiambo B, Ngure K, Ronen K, Sharma M, John-Stewart G, Richardson B, Stern J, Unger J, Udren J, Watoyi S, Pintye J, Kinuthia J. A Text Messaging-Based Support Intervention to Enhance Pre-exposure Prophylaxis for HIV Prevention Adherence During Pregnancy and Breastfeeding: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 30;12:e41170. doi: 10.2196/41170. PMID 36716092